CLINICAL TRIAL: NCT04856410
Title: Temporal Nature of Cognitive and Visuospatial Brain Domain Changes During Long-Duration Low-Earth Orbit Missions (Spatial Cognition)
Brief Title: Effects of Long-Duration Spaceflight on General and Spatial Cognition and Its Neural Basis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); DLR German Aerospace Center (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Mathias Basner, MD, PhD, Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 843851; 80NSSC19K1046 (Other Grant/Funding Number: National Aeronautics and Space Administration (NASA)); 50WB2115 (Other Grant/Funding Number: German Aerospace Center (DLR))
Record Dates: First submitted 2021-02-25; First posted 2021-04-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Brain Structure; Cognitive Performance
Keywords: Astronauts; Spaceflight; Cognition; Long Duration Spaceflight
MeSH Terms: interventions — Space Flight

STUDY DESIGN:
Intervention Model Description: This study will investigate 5 astronauts on 6-month ISS missions, 2 astronauts on 12-month ISS missions, and 7 control subjects that are matched to astronauts and investigated at similar time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 6-Month Arm (Experimental): Astronauts on 6-month International Space Station missions will be exposed to spaceflight for a duration of 6 months. Biometric and cognitive data will routinely be collected.
  Interventions: Other: Spaceflight
- 12-Month Arm (Experimental): Astronauts on 12-month International Space Station missions will be exposed to spaceflight for a duration of 12 months. Biometric and cognitive data will routinely be collected.
  Interventions: Other: Spaceflight
- No Intervention (Experimental): Subjects matched to 12-month astronauts that stay on Earth and are investigated at similar time points.
  Interventions: Other: Controls

INTERVENTIONS:
Other: Spaceflight — Exposure to the spaceflight environment on the International Space Station for 2, 6, or 12 months.
  Arms: 12-Month Arm; 6-Month Arm
Other: Controls — No intervention
  Arms: No Intervention

SUMMARY:
This study investigates the effects of extended-duration spaceflight (12-month International Space Station missions) on general cognitive performance (measured with the Cognition test battery), spatial cognition, structural and functional brain changes in general, and hippocampal plasticity more specifically relative to the shorter 6-month and 2-month missions.

DETAILED DESCRIPTION:
This is an international proposal consisting of two projects with synergistic aims that will be carried out in a joint effort by the National Aeronautics and Space Administration (NASA) and the German Aerospace Center (DLR) as well as the European Space Agency (ESA). The project targets NASA's particular interest in studying the 'Cognitive-perceptual-visuospatial brain domain changes due to isolation and confinement' as part of the Complement of Integrated Protocols for Human Exploration Research (CIPHER) project on the International Space Station (ISS). The collected data will demonstrate whether prolonging mission duration to one year will have detrimental effects on general cognitive performance (measured with the Cognition test battery), spatial cognition, structural and functional brain changes in general, and hippocampal plasticity more specifically relative to the shorter 6-month and 2-month ISS missions. Using state-of-the-art neuroimaging techniques, investigators will determine the biological basis for any changes in cognitive performance, with a focus on hippocampal plasticity and spatial cognition. Similar data already gathered on the ISS and in several short- and long-duration space analog environments will be used to generate a normative data base for long-duration missions. Finally, investigators will derive dose-response relationships between cognitive-visuospatial brain domain changes and mission duration that will allow predicting vulnerability to adverse cognitive or behavioral impairment and psychiatric disorders on interplanetary expeditions such as a mission to Mars. The two projects will deliver a highly unique and comprehensive set of integrated neuroimaging and neurocognitive tools for the evaluation and ultimately prevention of adverse effects on brain structure and function that lead to behavioral effects associated with exploration-type missions.

ELIGIBILITY:
Inclusion Criteria:

1. Astronauts (according to NASA requirements)
2. Normal, healthy volunteers (astronaut surrogates) - Astronaut surrogates will be matched for sex, age and education relative to astronauts

Exclusion Criteria:

For astronauts and normal, healthy volunteers (astronaut surrogates):

1. Subjects that do not comply with the MRI testing requirements. The following and other conditions may exclude the subject from MRI scanning or require additional examination to assess specific contraindications:

   * Tinnitus;
   * Sensori-neural hearing loss > 30 decibels (dB);
   * Pace-maker or internal defibrillator;
   * metallic implants (e.g. orthopedic plates after bone fractures, joint replacements, surgical staples or clips, artificial heart valves, stents, cava filters);
   * Metallic splinters (e.g. after an accident or due to war injury);
   * Non-removable dental brace;
   * Intrauterine contraceptive devices (IUD) that are not MRI-compatible;
   * Cochlear implant (implanted hearing device);
   * Medication pump;
   * Acupuncture needle;
   * Other foreign bodies/objects which are non-removable;
   * Pregnancy (or its possibility);
   * Previous brain and/or heart surgery.
   * Tattoos and/or permanent make-up in the body (some inks contain metallic particles).
2. Female subjects in this study are either astronauts or will model those in the astronaut population for whom participation in space missions is not allowed during pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive performance | Change from pre-flight performance (average of tests performed 180, 120 and 60 days prior to launch) to in-flight performance (average of all tests: 1 month mission = 1 test, 2 months = 2 tests, 6 months = 6 tests, 12 months = 12 tests)
  Cognitive efficiency across domains as determined with the Cognition test battery
Local task activation Cognition | Change from pre-flight local task activation (investigated 60 days prior to launch) to post-flight local task activation (investigated 5 days and 30 days after return to Earth)
  fMRI local task activation while performing the MRI version of Cognition in the scanner
Spatial cognition performance | Change from pre-flight performance (average of tests performed 180, 120 and 60 days prior to launch) to in-flight performance (average of all tests: 1 month mission = 1 test, 2 months = 2 tests, 6 months = 4 tests, 12 months = 7 tests)
  Accuracy and reaction times for each cognitive task as determined with the Spatial Cognition test batteries
Structural brain changes | Change from pre-flight local task activation (investigated 60 days prior to launch) to post-flight (investigated 5 days and 30 days after return to Earth)
  Structural brain changes assessed with MRI
Local task activation Spatial Cognition | Change from pre-flight local task activation (investigated 60 days prior to launch) to post-flight local task activation (investigated 5 days and 30 days after return to Earth)
  fMRI local task activation while performing visuospatial tasks in the scanner
Brain-Derived Neurotropic Factor (BDNF) | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Brain-Derived Neurotropic Factor (BDNF)

SECONDARY OUTCOMES:
Insulin-like Growth Factor 1 (IGF-1) | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Insulin-like Growth Factor 1 (IGF-1)
Vascular Endothelial Growth Factor (VEGF) | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Vascular Endothelial Growth Factor (VEGF)
Oxytocin | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Oxytocin
Interleukin (IL)-1 | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Interleukin (IL)-1
Interleukin (IL)-1ra | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Interleukin (IL)-1ra
Interleukin (IL)-10 | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Interleukin (IL)-10
Tumor Necrosis Factor a (TNFa) | Change from pre-flight values (average of blood drawn180 and 60 days prior to launch) to in-flight values (average of all in-flight blood draws: 1 month mission = 1 draw, 2 months = 2 draws, 6 months = 4 draws,12 months = 7 draws)
  Changes in Tumor Necrosis Factor a (TNFa)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Johnson Space Center (JSC), Houston, Texas
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
There will only be data sharing within our research group (CIPHER).

REFERENCES:
- [Background] Basner M, Moore TM, Hermosillo E, Nasrini J, Dinges DF, Gur RC, Johannes B. Cognition Test Battery Performance Is Associated with Simulated 6df Spacecraft Docking Performance. Aerosp Med Hum Perform. 2020 Nov 1;91(11):861-867. doi: 10.3357/AMHP.5602.2020. PMID 33334406
- [Background] Afshinnekoo E, Scott RT, MacKay MJ, Pariset E, Cekanaviciute E, Barker R, Gilroy S, Hassane D, Smith SM, Zwart SR, Nelman-Gonzalez M, Crucian BE, Ponomarev SA, Orlov OI, Shiba D, Muratani M, Yamamoto M, Richards SE, Vaishampayan PA, Meydan C, Foox J, Myrrhe J, Istasse E, Singh N, Venkateswaran K, Keune JA, Ray HE, Basner M, Miller J, Vitaterna MH, Taylor DM, Wallace D, Rubins K, Bailey SM, Grabham P, Costes SV, Mason CE, Beheshti A. Fundamental Biological Features of Spaceflight: Advancing the Field to Enable Deep-Space Exploration. Cell. 2020 Nov 25;183(5):1162-1184. doi: 10.1016/j.cell.2020.10.050. PMID 33242416
- [Background] Basner M, Hermosillo E, Nasrini J, Saxena S, Dinges DF, Moore TM, Gur RC. Cognition test battery: Adjusting for practice and stimulus set effects for varying administration intervals in high performing individuals. J Clin Exp Neuropsychol. 2020 Jul;42(5):516-529. doi: 10.1080/13803395.2020.1773765. Epub 2020 Jun 15. PMID 32539487
- [Background] Nasrini J, Hermosillo E, Dinges DF, Moore TM, Gur RC, Basner M. Cognitive Performance During Confinement and Sleep Restriction in NASA's Human Exploration Research Analog (HERA). Front Physiol. 2020 Apr 28;11:394. doi: 10.3389/fphys.2020.00394. eCollection 2020. PMID 32411017
- [Background] Lee G, Moore TM, Basner M, Nasrini J, Roalf DR, Ruparel K, Port AM, Dinges DF, Gur RC. Age, Sex, and Repeated Measures Effects on NASA's "Cognition" Test Battery in STEM Educated Adults. Aerosp Med Hum Perform. 2020 Jan 1;91(1):18-25. doi: 10.3357/AMHP.5485.2020. PMID 31852569
- [Background] Scully RR, Basner M, Nasrini J, Lam CW, Hermosillo E, Gur RC, Moore T, Alexander DJ, Satish U, Ryder VE. Effects of acute exposures to carbon dioxide on decision making and cognition in astronaut-like subjects. NPJ Microgravity. 2019 Jun 19;5:17. doi: 10.1038/s41526-019-0071-6. eCollection 2019. PMID 31240239
- [Background] Garrett-Bakelman FE, Darshi M, Green SJ, Gur RC, Lin L, Macias BR, McKenna MJ, Meydan C, Mishra T, Nasrini J, Piening BD, Rizzardi LF, Sharma K, Siamwala JH, Taylor L, Vitaterna MH, Afkarian M, Afshinnekoo E, Ahadi S, Ambati A, Arya M, Bezdan D, Callahan CM, Chen S, Choi AMK, Chlipala GE, Contrepois K, Covington M, Crucian BE, De Vivo I, Dinges DF, Ebert DJ, Feinberg JI, Gandara JA, George KA, Goutsias J, Grills GS, Hargens AR, Heer M, Hillary RP, Hoofnagle AN, Hook VYH, Jenkinson G, Jiang P, Keshavarzian A, Laurie SS, Lee-McMullen B, Lumpkins SB, MacKay M, Maienschein-Cline MG, Melnick AM, Moore TM, Nakahira K, Patel HH, Pietrzyk R, Rao V, Saito R, Salins DN, Schilling JM, Sears DD, Sheridan CK, Stenger MB, Tryggvadottir R, Urban AE, Vaisar T, Van Espen B, Zhang J, Ziegler MG, Zwart SR, Charles JB, Kundrot CE, Scott GBI, Bailey SM, Basner M, Feinberg AP, Lee SMC, Mason CE, Mignot E, Rana BK, Smith SM, Snyder MP, Turek FW. The NASA Twins Study: A multidimensional analysis of a year-long human spaceflight. Science. 2019 Apr 12;364(6436):eaau8650. doi: 10.1126/science.aau8650. PMID 30975860
- [Background] Basner M, Nasrini J, Hermosillo E, McGuire S, Dinges DF, Moore TM, Gur RC, Rittweger J, Mulder E, Wittkowski M, Donoviel D, Stevens B, Bershad EM; SPACECOT Investigator Group. Effects of -12 degrees head-down tilt with and without elevated levels of CO2 on cognitive performance: the SPACECOT study. J Appl Physiol (1985). 2018 Mar 1;124(3):750-760. doi: 10.1152/japplphysiol.00855.2017. Epub 2017 Dec 14. PMID 29357516
- [Background] Moore TM, Basner M, Nasrini J, Hermosillo E, Kabadi S, Roalf DR, McGuire S, Ecker AJ, Ruparel K, Port AM, Jackson CT, Dinges DF, Gur RC. Validation of the Cognition Test Battery for Spaceflight in a Sample of Highly Educated Adults. Aerosp Med Hum Perform. 2017 Oct 1;88(10):937-946. doi: 10.3357/AMHP.4801.2017. PMID 28923143
- [Background] Basner M, Savitt A, Moore TM, Port AM, McGuire S, Ecker AJ, Nasrini J, Mollicone DJ, Mott CM, McCann T, Dinges DF, Gur RC. Development and Validation of the Cognition Test Battery for Spaceflight. Aerosp Med Hum Perform. 2015 Nov;86(11):942-52. doi: 10.3357/AMHP.4343.2015. PMID 26564759
- [Background] Basner M, Dinges DF, Mollicone DJ, Savelev I, Ecker AJ, Di Antonio A, Jones CW, Hyder EC, Kan K, Morukov BV, Sutton JP. Psychological and behavioral changes during confinement in a 520-day simulated interplanetary mission to mars. PLoS One. 2014 Mar 27;9(3):e93298. doi: 10.1371/journal.pone.0093298. eCollection 2014. PMID 24675720
- [Background] Basner M, Dinges DF, Mollicone D, Ecker A, Jones CW, Hyder EC, Di Antonio A, Savelev I, Kan K, Goel N, Morukov BV, Sutton JP. Mars 520-d mission simulation reveals protracted crew hypokinesis and alterations of sleep duration and timing. Proc Natl Acad Sci U S A. 2013 Feb 12;110(7):2635-40. doi: 10.1073/pnas.1212646110. Epub 2013 Jan 7. PMID 23297197
- [Background] Mendt S, Gunga HC, Felsenberg D, Belavy DL, Steinach M, Stahn AC. Regular exercise counteracts circadian shifts in core body temperature during long-duration bed rest. NPJ Microgravity. 2021 Jan 5;7(1):1. doi: 10.1038/s41526-020-00129-1. PMID 33402671
- [Background] Chouker A, Stahn AC. COVID-19-The largest isolation study in history: the value of shared learnings from spaceflight analogs. NPJ Microgravity. 2020 Oct 22;6:32. doi: 10.1038/s41526-020-00122-8. eCollection 2020. PMID 33110938
- [Background] Friedl-Werner A, Brauns K, Gunga HC, Kuhn S, Stahn AC. Exercise-induced changes in brain activity during memory encoding and retrieval after long-term bed rest. Neuroimage. 2020 Dec;223:117359. doi: 10.1016/j.neuroimage.2020.117359. Epub 2020 Sep 10. PMID 32919056
- [Background] Roberts DR, Stahn AC, Seidler RD, Wuyts FL. Towards understanding the effects of spaceflight on the brain. Lancet Neurol. 2020 Oct;19(10):808. doi: 10.1016/S1474-4422(20)30304-5. Epub 2020 Sep 16. No abstract available. PMID 32949538
- [Background] Maggioni MA, Merati G, Castiglioni P, Mendt S, Gunga HC, Stahn AC. Reduced vagal modulations of heart rate during overwintering in Antarctica. Sci Rep. 2020 Dec 11;10(1):21810. doi: 10.1038/s41598-020-78722-3. PMID 33311648
- [Background] Stahn AC, Riemer M, Wolbers T, Werner A, Brauns K, Besnard S, Denise P, Kuhn S, Gunga HC. Spatial Updating Depends on Gravity. Front Neural Circuits. 2020 Jun 5;14:20. doi: 10.3389/fncir.2020.00020. eCollection 2020. PMID 32581724
- [Background] Stahn AC, Gunga HC, Kohlberg E, Gallinat J, Dinges DF, Kuhn S. Brain Changes in Response to Long Antarctic Expeditions. N Engl J Med. 2019 Dec 5;381(23):2273-2275. doi: 10.1056/NEJMc1904905. No abstract available. PMID 31800997
- [Background] Stahn AC, Werner A, Opatz O, Maggioni MA, Steinach M, von Ahlefeld VW, Moore A, Crucian BE, Smith SM, Zwart SR, Schlabs T, Mendt S, Trippel T, Koralewski E, Koch J, Chouker A, Reitz G, Shang P, Rocker L, Kirsch KA, Gunga HC. Increased core body temperature in astronauts during long-duration space missions. Sci Rep. 2017 Nov 23;7(1):16180. doi: 10.1038/s41598-017-15560-w. PMID 29170507
- [Background] Strewe C, Moser D, Buchheim JI, Gunga HC, Stahn A, Crucian BE, Fiedel B, Bauer H, Gossmann-Lang P, Thieme D, Kohlberg E, Chouker A, Feuerecker M. Sex differences in stress and immune responses during confinement in Antarctica. Biol Sex Differ. 2019 Apr 16;10(1):20. doi: 10.1186/s13293-019-0231-0. PMID 30992051
- See also: Reference article that does not have a pubmed ID yet "Head-Down Tilt Position, but Not the Duration of Bed Rest Affects Resting State Electrocortical Activity" — https://www.frontiersin.org/articles/10.3389/fphys.2021.638669/full

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT04856410/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04856410/ICF_001.pdf